CLINICAL TRIAL: NCT07045597
Title: Intranasal Midazolam for Preanasthetic Sedation for Preschool Children Undergoing Adenotonsillectomy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ramadan Hassan, Resident, Department of Anesthesia, Intensive Care and Pain management, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-3-08MS
Record Dates: First submitted 2025-06-14; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Adenotonsillar Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal normal saline for preanasthetic sedation for Adenotonsillectomy (Placebo Comparator): Patient will receive intranasal normal saline equivalent volume who take midazolam intranasal by dose 1 ml saline by insulin syringe as a control group
  Interventions: Drug: intranasal normal saline for preanasthetic sedation for Adenotonsillectomy
- intranasal midazolam for preanasthetic sedation for Adenotonsillectomy (Active Comparator): Patient will receive intranasal midazolam by dose 0.2 mg/kg
  Interventions: Drug: intranasal midazolam for preanasthetic sedation for Adenotonsillectomy

INTERVENTIONS:
Drug: intranasal normal saline for preanasthetic sedation for Adenotonsillectomy — preschool children that will undergo adenotonsillectomy will receive intranasal normal saline equivalent volume who take midazolam intranasal by dose 1 ml saline by insulin syringe as a control group
  Arms: intranasal normal saline for preanasthetic sedation for Adenotonsillectomy
Drug: intranasal midazolam for preanasthetic sedation for Adenotonsillectomy — preschool children that will undergo adenotonsillectomy will receive intranasal midazolam by dose 0.2 mg/kg
  Arms: intranasal midazolam for preanasthetic sedation for Adenotonsillectomy

SUMMARY:
This study aims to evaluate the effectiveness of Intranasal Midazolam as preanasthetic sedation for preschool children (2-6)y undergoing adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patient of age 2-6 y
* ASA I-II children
* child scheduled for elective adenoidectomy , tonsillectomy and adenotonsillectomy

Exclusion Criteria:

* Parent refusal .
* Allergy to any of the drug included in this study
* Nasal infection , allergy and pathology
* Mentally affected children , neurological disable .
* Blood disesases and any other contraindications of surgery

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
sedative effect of preanesthetic Midazolam | 5 minutes,10 minutes and 15 minutes preoperative
  Glasgow coma scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Korsch BM. The child and the operating room. Anesthesiology. 1975 Aug;43(2):251-7. doi: 10.1097/00000542-197508000-00010. No abstract available. PMID 1098522
- [Background] Rochette A, Julia JM, Evrard O, Ricard C, Jullien Y, Du Cailar J. [Intramuscular premedication with midazolam in infants and children]. Ann Fr Anesth Reanim. 1984;3(5):346-50. doi: 10.1016/s0750-7658(84)80071-4. French. PMID 6497079
- [Background] Rita L, Seleny FL, Mazurek A, Rabins SY. Intramuscular midazolam for pediatric preanesthetic sedation: a double-blind controlled study with morphine. Anesthesiology. 1985 Nov;63(5):528-31. doi: 10.1097/00000542-198511000-00009. No abstract available. PMID 2932039